CLINICAL TRIAL: NCT07335146
Title: Modélisation de l'œil Myope Infantile Par IRM et OCT
Brief Title: Eye Imaging for the Study of Childhood Myopia
Acronym: SELENA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WS10445; 2025-A00844-45 (Registry Identifier: ANSM RCB)
Record Dates: First submitted 2026-01-05; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hyperopia and Myopia
Keywords: myopia; eye anatomy; ophthalmological measurements
MeSH Terms: conditions — Hyperopia; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI and ophthalmological measurements (Experimental): All enrolled participants will undergo the same eye examinations such as head MRI and ophthalmological measurements
  Interventions: Device: Ophtalmic measurements to estimate geometrical distances; Device: MRI; Device: Ophtalmic measurements to measure wavefront aberrations

INTERVENTIONS:
Device: Ophtalmic measurements to estimate geometrical distances — Patients will undergo routine ophthalmic examinations, such as ocular biometry to estimate axial length and corneal topography. Anatomical characteristics will then be derived from the geometric measurements obtained from each device. All measurements are non-invasive and non-ionizing. They all involve conventional ophthalmic devices that are widely used in clinical settings.
Device: MRI — Participants will undergo Magnetic Resonance Imaging (MRI) to image their eyes. A head antenna will be used. All measurements are non-invasive.
Device: Ophtalmic measurements to measure wavefront aberrations — Patients will undergo ophthalmic measurements to assess ocular wavefront aberrations. These measurements will be performed using commercially available devices that are widely accepted in routine clinical practice. All procedures are non-invasive and non-ionizing.

SUMMARY:
Myopia (nearsightedness) is increasing worldwide and is becoming a serious public health problem. Studies estimate that by 2050, if no action is taken, almost half of the world's population will be myopic. About 10% of people could develop severe myopia, which increases the risk of serious eye problems such as retinal detachment, damage to the macula, or glaucoma.

Children are particularly affected because myopia often worsens as they grow. Several treatments are now available to slow the progression of myopia in children, but these treatments are not equally effective for everyone. Some children respond better than others, and the reasons for these differences are not yet well understood. One possible explanation is that differences in eye anatomy may influence the effectiveness of a treatment. This suggests that myopia treatments may need to be tailored to each child. By studying the anatomy of the eye, researchers could improve and personalize myopia control strategies.

The study entitled "Eye imaging for the study of childhood myopia" aims to better understand the structure of children's eyes. The study will collect clinical data, including images of the eye taken with MRI and measurements of the eye obtained using standard eye examination devices. The data will then be analyzed using image-processing and statistical methods to allow a detailed study of children's eye anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Spherical equivalent under cycloplegia greater -6.5 D and less than 2 D
* Beneficiary of social security
* Written consent from both holders of parental authority (or from one in case of exclusive parental authority)

Exclusion Criteria:

* Declared neurological deficit, including history of epileptic pathology or sensory-motor coordination disorders, vestibular or cerebellar pathology (for example, balance disorders)
* Current or progressive pathology of the eyes or their appendages that may affect vision, other than myopia (examples: glaucoma, retinitis pigmentosa…)
* Declared aphakia or pseudophakia (intraocular implant)
* Ocular motility problem such as strabismus or nystagmus
* Contraindication to MRI (claustrophobia, implanted devices such as pacemaker, etc.)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Eye anatomy | From enrollment to 3 months after enrollment
  This set of data will enable an in-depth study of the eye anatomy: MRI will provide anatomical characteristics of the eyeball and its surrounding tissues such as the optical nerve. Ophtalmic measurements will provide anatomical characteristics of the eye's refractive system, such as corneal pachymetry, with optimal geometric resolution. Thus, MRI images and ophtalmic measurements will be combined to study the overall eye anatomy.
  Period: From inclusion up to 3 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because participant consent did not include permission for data sharing.